CLINICAL TRIAL: NCT06855797
Title: Characterization of Chronic Pain in Elderly Population with Emphasis on Differences Between Gender
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 43535915.0.0000.0068
Record Dates: First submitted 2017-07-10; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2017-07

CONDITIONS: Elderly; Chronic Pain; Gender
MeSH Terms: conditions — Chronic Pain; Coitus | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Male: Male, patients
  Interventions: Other: Observation
- Female: Female patients
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — questionnaire

SUMMARY:
Introduction: It is estimated that by 2025 there will be approximately 1.2 billion people above 60 years old. Global projections indicate that by 2050 there will be about 2 billion elders, 80% of them living in developing countries. Researches on the relationship between pain and aging are currently much valued within the health sciences, the ultimate goal being the provision of adequate pain control for the growing number of elders in society. Objectives: To characterize chronic pain in the elderly population and evaluate pain threshold to mechanical stimulation, with emphasis on gender differences. Methods: This study refers to a cross-sectional study to be conducted in convenience samples of a primary care unit (Geraldo Horacio de Paula Souza) that follows elders and the Department of Geriatrics of the university hospital of the School of Medicine of Universidade de São Paulo (Hospital das Clínicas). At least 200 participants of each gender, aged 65 or above, will be selected to participate. Chronic pain will be that lasting for six or more months (either continuous or recurrent, as recommended by the International Association For the Study of Pain). Participants will be searched about their demographic and socioeconomic backgrounds, and asked to answer the following questionnaires: the Mini Mental State Examination, a structured questionnaire for activities of daily living, a structured questionnaire for instrumental activities of daily living, Beck Anxiety Inventory, Geriatric Depression Scale, the five dimensions European Quality of Life assessment (EQ5D) and Brief Pain Inventory. Participants will also be evaluated regarding pain threshold to mechanical stimuli using algometer. Descriptive statistics of the sample will be displayed as means, medians, standard deviations and proportions. For testing for differences between males and females, a significance level of 5% will be used. Keywords: elderly, chronic pain, gender.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the geriatrics clinic at the Central Institute (IC) of the Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HCFMUSP) or the Geraldo Horácio de Paula Souza School of Public Health Center of the University of São Paulo
* Be over 65 years old
* Accept study participation
* Have read, understood, agreed and signed the TCLE

Exclusion Criteria:

* Cognitive difficulty in understanding and responding to research questions
* Do not accept participation in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self representation
Study Population: Patient of the geriatrics clinic at the Central Institute (IC) of the Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HCFMUSP) or the Geraldo Horácio de Paula Souza School of Public Health Center of the University of São Paulo
Sampling Method: Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity to pressure pain 5 minutes post recruitment | applied minutes 5 after recruitment of the subject.
  Pain evaluation throught algometer 5 minutes post recruitment
Sensitivity to pressure pain 10 minutes post recruitment | applied minutes 10 after recruitment of the subject.
  Pain evaluation throught algometer 10 minutes post recruitment
Sensitivity to pressure pain 15 minutes post recruitment | applied minutes 15 after recruitment of the subject.
  Pain evaluation throught algometer 15 minutes post recruitment

SECONDARY OUTCOMES:
Mini Mental State Examination | applied in beginning of the interview
  Mental state evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valkenburg HA. Epidemiologic considerations of the geriatric population. Gerontology. 1988;34 Suppl 1:2-10. doi: 10.1159/000212980. PMID 3266492
- [Background] Chesterton LS, Barlas P, Foster NE, Baxter DG, Wright CC. Gender differences in pressure pain threshold in healthy humans. Pain. 2003 Feb;101(3):259-266. doi: 10.1016/S0304-3959(02)00330-5. PMID 12583868
- [Background] Riley JL 3rd, Robinson ME, Wise EA, Myers CD, Fillingim RB. Sex differences in the perception of noxious experimental stimuli: a meta-analysis. Pain. 1998 Feb;74(2-3):181-7. doi: 10.1016/s0304-3959(97)00199-1. PMID 9520232
- [Background] Bartley EJ, Fillingim RB. Sex differences in pain: a brief review of clinical and experimental findings. Br J Anaesth. 2013 Jul;111(1):52-8. doi: 10.1093/bja/aet127. PMID 23794645
- [Background] Peat G, Thomas E, Handy J, Croft P. Social networks and pain interference with daily activities in middle and old age. Pain. 2004 Dec;112(3):397-405. doi: 10.1016/j.pain.2004.09.029. PMID 15561396